CLINICAL TRIAL: NCT01114698
Title: A Randomized, Double-Blind, Parallel Group, Active- and Placebo-Controlled Study to Assess the Efficacy and Safety of JNJ26489112 in Adult Subjects With Treatment-Resistant Major Depressive Disorder
Brief Title: A Safety and Efficacy Study of JNJ26489112 in Patients With Treatment-Resistant Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to sponsor portfolio decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR016579; 26489112MDD2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-04-22; First posted 2010-05-03 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder; Venlafaxine XR (EFFEXOR XR); 26489112; JNJ26489112
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — N-((6-chloro-2,3-dihydrobenzo(1,4)dioxin-2-yl)methyl)sulfamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- JNJ26489112 (Experimental)
  Interventions: Drug: JNJ26489112
- Venlafaxine XR (Active Comparator)
  Interventions: Drug: Venlafaxine XR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine XR — Venlafaxine XR 75 mg/day administered orally once daily as 2 capsules identical in appearance to JNJ26489112 during the first week increased to 150 mg/day during weeks 2 through 6.
  Arms: Venlafaxine XR
Drug: Placebo — Placebo: 2 capsules identical in appearance to JNJ26489112 and venlafaxine XR orally administered once daily for 6 weeks.
  Arms: Placebo
Drug: JNJ26489112 — JNJ26489112 500 mg/day orally administered once daily as 2 capsules for the first 3 weeks, then dose may be increased to 1000 mg/day by week 4.
  Arms: JNJ26489112

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of JNJ26489112 compared with an active control (Venlafaxine XR) and placebo in patients with Treatment-Resistant Major Depressive Disorder.

DETAILED DESCRIPTION:
This is a randomized (patients assigned to treatment groups by chance), double-blind (neither the study physician nor the patient will know the identification of treatment assigned), active- and placebo-controlled study to assess the efficacy and safety of JNJ26489112 in adult patients with treatment-resistant major depressive disorder (MDD). The active control used in the study is venlafaxine extended-release [XR], an antidepressant drug used to treat patients with MDD. A target of 150 patients will be randomly assigned (like flipping a coin) to 1 of 3 treatment groups with approximately 50 patients planned per treatment group. This study consists of a screening phase of up to 4 weeks, a 6-week double-blind treatment phase, and a safety follow-up period that includes a 1-week taper phase (described below). During the screening phase, patients who meet entry criteria for the study will be tapered off their current psychotropic medications (medications affecting the mind or mood or other mental processes) prior to randomization in the double-blind treatment phase of the study. In the double-blind treatment phase, patients will be randomly assigned to receive either 2 capsules of JNJ26489112, venlafaxine XR (the active comparator), or placebo (a sugar pill) once daily for 6 weeks. Upon completion of the double-blind treatment phase or when patients discontinue study drug at any time point during the double-blind treatment phase, study medication will be tapered and/or discontinued in a blinded manner over a 1-week period. A Data Monitoring Committee (DMC) made up of individuals not involved in the conduct of the study will monitor safety during the study. The primary outcome measure will be the change from baseline to end point (after 6 weeks of treatment or at the time of early withdrawal from the study) in the total score from the Montgomery-Asberg Depression Rating Scale (MADRS, a scale that physicians use to measure the severity of depression in patients and changes in depression due to antidepressant treatment). Patient safety will be monitored during the study by evaluating adverse events (side effects) reported and findings from clinical laboratory test results, 12-lead electrocardiograms (ECGs), vital sign measurements, body weight measurements and physical, neurologic, and ophthalmologic examinations performed. Blood samples for assessing pre- and post dose levels of JNJ26489112 or venlafaxine will be obtained at protocol-specified time points during the study. In addition, a blood sample will be obtained from all enrolled patients at Visit 2 for pharmacogenomics research (research to help identify genetic markers of response, to explain variability in the data, or to address emerging clinical issues). Patients will receive double-blind treatment with 2 capsules of JNJ26489112 (500 mg/day during the first 3 weeks that may be increased up to 1000 mg/day by week 4), venlafaxine XR (75 mg/day during week 1 increased to 150 mg/day during weeks 2-6]), or placebo orally (by mouth) with food once daily for 6 weeks. After 6 weeks, venlafaxine XR 150 mg/day will be tapered to one 75 mg/day capsule for 1 week and patients receiving JNJ26489112 or placebo will be switched to 1 capsule of placebo for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revised (DMS-IV-TR) criteria for diagnosis of moderate or severe major depression without psychotic features
* Have a score >=40 on the subject-rated Inventory of Depressive Symptoms-Self-Report - 30-item (IDS-SR30) At Screening (Visit 1) and Randomization (Visit 2)
* Have a history of inadequate treatment response (as defined by failure to improve with a trial of adequate dosage and duration) with 2 antidepressants during the current episode, but no more than 4 antidepressant failures for lifetime
* Be in good general health prior to study participation with no clinically relevant abnormalities as assessed by the investigator and determined by: medical history, physical examination, blood chemistry, hematology, urinalysis, and electrocardiogram (ECG)
* Be within a body mass index (BMI) of >=18 and <35 kg/m2 at Screening (Visit 1)

Exclusion Criteria:

* Have a DSM-IV diagnosis of current (active) generalized anxiety disorder, panic disorder, obsessive compulsive disorder, posttraumatic stress disorder, anorexia nervosa, or bulimia nervosa
* Have a history or current diagnosis of a psychotic disorder, bipolar disorder, mental retardation, or borderline personality disorders, mood disorder with postpartum onset, somatoform disorders, chronic fatigue syndrome or fibromyalgia
* Have a history of previous non-response to an adequate treatment with venlafaxine XR (defined as >=6 weeks of 75 to 150 mg/day or more)
* Have documented disease of the central nervous system that could interfere with the study assessments (including but not limited to: stroke, tumor, multiple sclerosis, Parkinson's disease, Alzheimer's disease, Huntington's disease, seizure disorder requiring current anticonvulsants, history of brain injury or trauma, or neurosyphilis)
* Have a history of alcohol or substance (except nicotine and caffeine) dependence or abuse according to DSM-IV criteria in the past 12 months prior to Screening
* Received an experimental drug or used an experimental medical device within 60 days before the planned start of treatment (Day 1) or have participated in 2 or more clinical studies in the previous 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (10 item diagnostic questionnaire measuring the severity of depression) | Baseline and 6 weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | At each weekly visit during the study (screening through completion of the study [Week 7])
Mean Change in Inventory of Depressive Symptoms (IDS) and Clinical Global Impression (CGI) | At Visits 1, 2, 4, 6, 8, and 9 (Screening, Baseline, Week 2, Week 4, Week 6, and Week 9)
Findings from ophthalmologic examinations | Before the first dose of study drug, at Week 3, and after the last dose in the double-blind phase of the study (Week 7 or at the time of early termination from the study)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- United States (14):
  - Arcadia, California
  - Escondido, California
  - San Diego, California
  - Hartford, Connecticut
  - Atlanta, Georgia
  - Naperville, Illinois
  - Brooklyn, New York
  - Garfield Heights, Ohio
  - Oklahoma City, Oklahoma
  - Dallas, Texas
  - Houston, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Middleton, Wisconsin